CLINICAL TRIAL: NCT03422705
Title: A Randomised, Placebo-controlled Pilot Trial to Examine the Efficacy of Interventions to Prevent Left Ventricular Remodelling in Patients Receiving New Pacemaker Implantation (OPT-Prevent-pilot).
Brief Title: A Pilot Study: Preventing Adverse Remodelling Following Pacemaker Implantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, KK Witte, Senior Lecturer in Cardiology, University of Leeds
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 242990
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Pacemakers, Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Lisinopril; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Sham Comparator): No intervention - no programming, no medical intervention.
  Interventions: Other: Standard care
- Optimised programming (Experimental): Optimised pacemaker programming to avoid right ventricular pacing.
  Interventions: Device: Optimised programming; Other: Standard care
- Medical therapy (Experimental): Lisinopril uptitrated to optimally tolerated dose.
  Interventions: Device: Optimised programming; Drug: Lisinopril; Other: Standard care

INTERVENTIONS:
Device: Optimised programming — Optimised programming to avoid RV pacing when possible.
  Arms: Medical therapy; Optimised programming
Drug: Lisinopril — Uptitration of lisinopril
  Arms: Medical therapy
Other: Standard care — No pacemaker adjustment or medical therapy

SUMMARY:
Almost 40,000 people in the United Kingdom receive a new pacemaker annually. Because the pacemaker does not use the heart's normal conduction system, electrical activity from the pacemaker spreads more slowly, disturbing the timing of the heart's contraction, which can lead to heart muscle weakness and heart failure (HF).

Those with the greatest requirement for a pacemaker and highest percentage of pacemaker beats are those at highest risk of heart muscle weakness.

This pilot study will be in two stages. Patients will be approached after their pacemaker implant. Allocation to all treatment arms will be at random.

At the normal 6w visit, all participants will undergo cardiac ultrasound, blood tests and complete a quality of life questionnaire. Participants will be allocated to optimal pacemaker programming (to limit pacemaker heartbeats) or standard care. Those allocated optimal programming will return 3m after the implant and those still needing a high proportion of pacemaker beats, will be asked to have a cardiac magnetic resonance (CMR) scan and will be randomly allocated to an angiotensin converting enzyme inhibitor (ACE inhibitor) a common treatment for blood pressure and HF or not. After another 6m all will undergo heart ultrasound, blood test and quality of life assessment, and where relevant, a second CMR scan.

DETAILED DESCRIPTION:
All patients booked for pacemaker clinic 6w following a new implant for heart block will receive an information sheet with their appointment letter. Potential participants will attend the National Institute of Health Research Clinical Research Facility at Leeds General Infirmary. Each participant will sign a consent form and undergo a baseline echocardiogram, a quality of life assessment (EQ5D-5L), and blood tests including B-type natriuretic peptide measurement. The investigators will record demographic and clinical variables including co-morbidities and current medication.

Patients will be allocated in a 1:2 allocation stratified for atrial rhythm (atrial fibrillation or sinus rhythm) to either standard care (sham programming) or intervention (protocolised pacing-avoidance programming. Patients will be called at 1w to ensure short term acceptability and safety and then reviewed at 3m after the implant. At that visit, a pacing check will establish the amount of RV pacing required. Those pacing >40% despite optimised programming will be asked to undergo a cardiac magnetic resonance (CMR) scan and will be randomly allocated to Lisinopril 5mg (ACEi) or no treatment. They will take one tablet daily and the dose will be increased 2 weekly to the maximally tolerated dose or 20mg daily. This will be supervised by the HF nurse. All patients will be reviewed at a further 6m (9m after their pacemaker procedure) with a repeat echocardiogram, blood test for BNP, QoL assessment, and those in phase two (lisinopril or not) will undergo a repeat CMR scan.

Choice of endpoints Left ventricular remodelling is a widely accepted surrogate endpoint in clinical studies, and therapy-related changes in LV structure and function are related morbidity/mortality outcomes. A 5% increase in mean LVEF was associated with an odds ratio (OR) of 0.86 [95%CI 0.77-0.96] for one-year mortality. LV end diastolic volume (LVEDV) also demonstrates a reliable link to mortality outcomes. A decrease of 10ml is associated with an OR of 0.95 [0.94-0.97] for one-year mortality, whilst a decrease in LV end systolic volume (LVESV) of 10ml is associated with an OR of 0.96 [0.93-0.98] for mortality at 1yr. The investigators will also measure change in indexed volumes such as LVESVi which is frequently used in pacemaker studies. A reduction in LVESVi of ≥15% is associated with better outcome in recipients of a CRT device.

Safety and patient tolerability The protocol of minimising unnecessary RV pacing was well tolerated. ACEi are well-tolerated with fewer than 15% of HF patients unable to tolerate any dose of short-acting enalapril. We expect a lower rate of discontinuation since patients will not have HF and lisinopril is longer-acting. In the Assessment of Treatment with Lisinopril and Survival study (ATLAS), there was adverse effect rate of 4.6% and symptomatic hypotension in 1%. Higher doses were associated with a greater effect, and the discontinuation rate was not related to dose. The investigators conservatively estimate that 10% patients will not tolerate ACEi.

Statistical considerations In estimating sample size, the investigators have followed the rules of thumb for pilot studies proposed by Browne to use at least 30 subjects, and the suggestions of Julious to include at least 12 subjects per treatment arm, and Teare et al for 70 subjects in total. The investigators have assumed that 20% will not have complete heart block at their 6w check, such that if they consent 75 patients, 60 will go through to randomisation, of whom 20 will be allocated standard care (group 1) and 40 will be randomly allocated to optimised pacing (group 2). Those in group 2 still pacing >40% in the RV, will be randomly allocated lisinopril or not in a 1:1 ratio. In addition to exploring the effects of an ACEi on pacing-induced remodelling using CMR in patients with no programming options, they will also be able to compare 6m remodelling in three groups using echocardiography: pacing <40% (n=25), pacing ≥40% (n=35), and pacing ≥40% but taking an ACEi (n=15).

Feasibility In Leeds, 35% of 450 patients receiving an RV pacemaker have heart block (n=160). Around 20% will be excluded due to an ejection fraction <45% (n=32) and a further 20% (n=26) will already be taking an ACE inhibitor. This leaves a pool of 100 people annually who might be eligible. An anonymised study log of people receiving a pacemaker for heart block but excluded for other reasons will be maintained until recruitment is completed.

Blinding The programming will be blinded but ACEi allocation will be open-label. Echocardiography and CMR scans will be performed/administered/reported by a blinded cardiac physiologist or CMR technician and physician. An unblinded cardiac physiologist will be available at each visit for programming questions.

Data analysis:

Statistical analysis plan The primary endpoint will be change in LVEF at 9m post-implant. Secondary outcomes will include other remodelling variables (LVEDV, LVESV), quality of life (EQ5D-5L), and estimated battery longevity at 9m. Patients will be analysed according to their randomised allocation and the difference between groups estimated using a general linear model adjusting for baseline LVEF. Analysis of other endpoints will use similar methods.

ELIGIBILITY:
Inclusion criteria:

* New RV pacemaker implant (<6 weeks)
* Willing and able to give informed consent
* Stable medical therapy (≥6w)

Exclusion criteria:

* Poor imaging quality
* Patients without heart block
* Guideline-mandated ACEi or ARB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | 6 months
  Difference in change between the groups

SECONDARY OUTCOMES:
Change in left ventricular end systolic diameter | 6 months
  Difference in change between the groups
Change in left ventricular end diastolic diameter | 6 months
  Difference in change between the groups

IPD SHARING:
Plan to Share IPD: No
This is just a pilot study